CLINICAL TRIAL: NCT02800447
Title: Procarbazine Hydrochloride Capsule (Natulan®) Clinical Trial Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zhaoke-NTL-2015-01
Record Dates: First submitted 2016-05-24; First posted 2016-06-15 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Advanced Hodgkin's Lymphoma
MeSH Terms: interventions — Procarbazine

ARMS (2):
- Treatment (Experimental): baseline BEACOPP regimen
  Interventions: Drug: Natulan
- controlled group (Active Comparator): ABVD regimen
  Interventions: Drug: ABVD

INTERVENTIONS:
Drug: Natulan — Each baseline BEACOPP regimen lasts 21 days, and each cycle consists of： Cyclophosphamide injection: 650mg/m2, IV infusion, day 1； Doxorubicin hydrochloride injection: 25mg/m2, IV infusion, day 1； Etoposide injection: 100mg/m2, IV infusion, day 1~3; Natulan (procarbazine hydrochloride capsule): 100mg/m2，po, day 1~7; Bleomycin hydrochloride injection: 10mg/m2, IV or IM, day 8; Vincristine: 1.4mg/m2 (single maximum dose is 2mg), IV infusion, day 8; Prednisone tablet: 40mg/m2, po, day 1~14
  Other Names: Procarbazine hydrochloride capsules
  Arms: Treatment
Drug: ABVD — Each ABVD cycle lasts 28 days1 cycle of the ABVD regimen consists of： Doxorubicin hydrochloride injection：25mg/m2，IV infusion，day 1 and 15; Dacarbazine injection：375mg/m2，IV infusion，day 1 and 15； Bleomycin injection：10mg/m2，IV or IM，day 1 and 15； Vincristine injection：1.4mg/m2 (single maximum dose is 2mg), IV infusion，day 1 and 15;
  Arms: controlled group

SUMMARY:
1. To observe and compare the overall response rate (ORR) of baseline BEACOPP and ABVD regimens for patients with advanced Hodgkin's lymphoma.
2. To evaluate the safety of Natulan® in Chinese patients with advanced Hodgkin's lymphoma

DETAILED DESCRIPTION:
This is a confirmatory open-label, randomized, controlled, multicenter study. Recruited subjects are to be randomized to treatment group and controlled group, with ratio of 1:1. Treatment group will accept baseline BEACOPP regimen, while controlled group will accept ABVD regimen.

The study design consisted of a screening phase of 1 week, a treatment phase of 24 or 32 weeks, and a post treatment follow-up of at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

* The subject is of age 18~65, both male and female;
* Newly pathologically diagnosed with classical Hodgkin's lymphoma (lymphocyte depletion type, lymphocyte rich type, nodular sclerosing type, and mixed cellularity type), who had not accepted previous treatment;
* Had stage IIB, III or IV disease, as assessed by the Ann Arbor classification;
* ECOG≤2, life expectancy ≥3 month;
* A negative serum pregnancy test required for sexually active women of childbearing potential;
* The subject voluntarily gives written informed consent to participate in the study.

Exclusion Criteria:

* Hematopoietic function:

  * Leukocyte <3,500/mm3（3.5×109/L）
  * Neutrophils <1,500/mm3（1.5×109/L）
  * Platelets <100,000/mm3（100×109/L）
* Intolerance to any of the active ingredients and/or excipients in the study medications;
* Severe central nervous system disorders and mental illness;
* Severe heart disease (congestive heart failure, uncontrolled hypertension, unstable coronary artery disease, or myocardial infarction, or severe arrhythmia). Echocardiography showed resting left ventricular ejection fraction (LVEF) < 50%);
* History of severe lung disease;
* AST or ALT>2.5×ULN，total bilirubin≥1.5×ULN，serum creatinine>1.5×ULN (for subject with liver metastases: AST or ALT>5xULN, total bilirubin ≥ 3xULN);
* Uncontrolled, systemic, active infection；
* Positive serology to HIV;
* HBsAg positive subjects can still be enrolled in the study, but researchers should follow "The consensus on the Treatment of Lymphoma with Hepatitis B Infections" to observe closely and/or provide prophylactic anti-HBV therapy (as per investigator's decision);
* Other previous or concomitant malignancy, except for basal cell carcinoma and/or cervical carcinoma in situ;
* The subject is receiving an investigational drug, or has participated in an investigational study within 30 days prior to screening;
* The subject is pregnant or lactating; or subjects of childbearing potential (both women and man subjects) do not want to take effective contraceptive measures during study period or within 3 months after study completes;
* Investigators believe subjects not suitable to participate in the study for other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | 45 months
  Compare the overall response rate (ORR) of baseline BEACOPP and ABVD regimens for in patients with advanced Hodgkin's lymphoma.

SECONDARY OUTCOMES:
safety as measured by changes of vital signs, ECG and AE number | 45 months